CLINICAL TRIAL: NCT00668590
Title: Improving Diabetes Care With Patient Decision Aids - A Randomized Controlled Trial in Community-based Primary Care
Brief Title: Improving Diabetes Care With Patient Decision Aids - A Trial in Community-based Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Robert Wood Johnson Foundation (Other); Foundation for Informed Medical Decision Making (Other)
Responsible Party: Dominick L. Frosch, Ph.D., Assistant Professor, UCLA Department of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: G08-01-038-01
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Patient video decision aid & telephone coaching
- 2 (Active Comparator)
  Interventions: Behavioral: Printed educational brochure

INTERVENTIONS:
Behavioral: Patient video decision aid & telephone coaching — The decision aid is a 30 minute video program that educates patients about their role in diabetes care. Telephone coaching will assist patients in initiating behavior change.
  Arms: 1
Behavioral: Printed educational brochure — The printed brochure is an educational brochure developed by the NIH.
  Arms: 2

SUMMARY:
Mounting evidence documents the positive impact of using patient decision aids (PtDA) to facilitate shared decision-making (SDM) between patients and physicians in preference sensitive contexts. But overall use of PtDAs across the broader US healthcare system remains low. More compelling evidence is needed to make the case for policies that would accelerate adoption of PtDAs in routine clinical practice in primary care settings that serve diverse and economically disadvantaged populations. The investigators believe that it is now time to move beyond the subjective evaluations of PtDAs that are commonly reported in clinical trials of PtDAs, to evaluate whether these tools can also change health behavior and improve health outcomes. Therefore, the investigators will build on their expertise in working with community-based physicians to evaluate a newly developed PtDA focused on diabetes, using a mixed-methods approach. The investigators patient sample will be drawn from primary care practices serving African American, Latino and Caucasian patients. The investigators will conduct a 2-group randomized controlled trial to evaluate the effects of the diabetes PtDA, combined with telephone coaching, in increasing patient self-care and self-efficacy, increasing diabetes knowledge and improving clinical measures including glycosylated hemoglobin A1c, lipids and blood pressure. The investigators will also explore variation in effects of the patient decision aid, comparing African American, Latino and Caucasian patients and conduct in-depth interviews with a randomly selected subset of trial participants to explore patient perceptions of the decision aid and variation across racial/ethnic groups. The investigators hypothesize that, compared to the control condition, participants assigned to receiving the video PtDA program and telephone coaching will report: greater self-efficacy and diabetes knowledge, more engagement in self-care behaviors, better glycemic control as measured by hemoglobin A1c, as well as lower quantitative LDL and blood pressure levels. The conceptual model guiding the investigators trial is the Integrative Model of Behavior Change. The model includes three primary determinants of behavior:

1. attitudes toward performing the behavior
2. perceived social norms about performing the behavior
3. self-efficacy. The investigators expect the diabetes PtDA to affect each of these constructs directly or indirectly.

ELIGIBILITY:
Inclusion Criteria:

1. At least 40 years old.
2. Diagnosed with Type 2 diabetes at least 1 year ago.
3. Attending the clinic for a routine diabetes follow-up visit.
4. Completed at least 2 clinic visits in the past 12 months.
5. Glycosylated hemoglobin A1c equal or greater than 8.0%
6. Owns a DVD player and television at home
7. Willing to provide informed consent.

Exclusion Criteria:

1. Primary language other than English.
2. Severe visual impairment
3. Currently enrolled in a diabetes education or support program, or participated in a diabetes education or support program in the last 6 months.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 6 months

SECONDARY OUTCOMES:
Diabetes self-care behaviors | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dominick L Frosch, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - UCLA Internal Medicine practices, Los Angeles, California
  - Community-based primary care practices, Los Angeles, California

REFERENCES:
- [Derived] Frosch DL, Uy V, Ochoa S, Mangione CM. Evaluation of a behavior support intervention for patients with poorly controlled diabetes. Arch Intern Med. 2011 Dec 12;171(22):2011-7. doi: 10.1001/archinternmed.2011.497. Epub 2011 Oct 10. PMID 21986347